CLINICAL TRIAL: NCT05926453
Title: Validation of Indirect Estimation Against Direct Gas Measurements of Cardiorespiratory Fitness Using the Modified Balke Protocol on a Treadmill in Patients With Spondylarthritis
Brief Title: Assessment of Cardiorespiratory Fitness in Spondylarthritis
Status: Active, not recruiting | Type: Observational
Sponsor: Diakonhjemmet Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DS-00772
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Spondylarthritis
Keywords: exercise test; validation study
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Maximal CPET: One maximal cardiopulmonary exercise test with simultaneous registration of direct gas measurements and the variables necessary for estimated cardiorespiratory fitness.
  Interventions: Other: Maximal cardiorespiratory exercise test

INTERVENTIONS:
Other: Maximal cardiorespiratory exercise test — previously described

SUMMARY:
Spondyloarthritis is a chronic inflammatory joint disease that affects the spine and sacroiliac joints. Most untreated patients eventually experience impaired mobility of the spine, pain and reduced physical function. Exercise is a cornerstone in the treatment of patients with spondylarthritis and it has been shown that high intensity exercise is just as effective in reducing disease activity as immunosuppressive medication. Additionally, patients with spondylarthritis have increased risk of cardiovascular disease both due to traditionally risk factors (obesity, high blood pressure etc) but also due to chronic inflammation. A maximal cardiopulmonary exercise test (CPET) is a measure of cardiorespiratory fitness that can be used to show progression of the exercise and which also is correlated to all-cause mortality and life expectancy.

The investigators will validate an indirect maximal CPET against the gold standard with direct gas exchange measurements in patients with spondylarthritis. The indirect test is less time consuming, requires less sophisticated equipment, has lesser requirements to test personnel and facilities, and has less expenditures than the direct test. With a validated indirect maximal CPET the test of cardiorespiratory fitness will be more accessible for patients with spondylarthritis both in-hospital but also municipal.

DETAILED DESCRIPTION:
Spondylarthritis (SpA) is a chronic inflammatory disease which affects sacroiliac joints, spine and peripheral joints with an onset usually before the age of 45 years. The prevalence is approximately 1.5% and correlated to the distribution of the genotype HLA-B27 in the population. Most untreated patients eventually experience limited mobility of the spine, pain, reduced physical function and fatigue. There is a considerable likelihood for significantly impaired quality-of-life, morbidity and work disability. Exercise is a cornerstone in the treatment of patients with SpA, and it has been shown that supervised high intensity interval training has equally positive effect on disease activity as biological immunomodulating treatment. The inflammatory joint diseases have a high prevalence of comorbidities such as cardiovascular disease (CVD) driven by both traditional and non-traditional risk factors. The CVDs are an important cause of premature mortality for patients with inflammatory joint diseases including SpA.. Traditional CVD risk factors such as obesity and lower levels of physical activity, coupled with non-traditional risk factors such as systemic inflammation, are key causal factors.

Cardiorespiratory fitness is a strong predictor of all-cause mortality and life expectancy also for patients with SpA, and improved cardiorespiratory fitness seems to reduce the risk of cardiovascular disease in a quantitative manner. The gold standard for measurement of an individual's cardiopulmonary fitness expressed as the peak oxygen consumption (VO2peak) is considered as the direct gas exchange measurements during maximal exercise of large muscle groups such as running, cycling, or swimming. However, the direct gas exchange measurement is time-consuming and requires technical instrumentation and highly skilled personnel, and it is therefore often more convenient to use estimates. For the maximal exercise test to measure correct VO2peak levels or estimate correct physical fitness the participants must be willing and capable of pushing themselves with the assistance of cheering from the technical personnel otherwise the VO2peak will be underestimated. It is therefore evident that the result of the performed test depends on the maximal effort being executed.

The modified Balke protocol is a protocol often used in maximal cardiopulmonary exercise testing (CPET) on a treadmill. According to this protocol the workload is increased by elevated inclination to a maximum of 15%. If the participant is capable of further increased workload the speed of the treadmill is increased till exhaustion of the participant. With the indirect test, VO2peak is estimated from the time to exhaustion (TTE), incline of the treadmill and the speed of the treadmill. The indirect test requires a treadmill with adjustable incline, heart rate monitor and a stopwatch. The direct VO2 measurement is performed with breath-by-breath gas exchange measurement of inspiratory and expiratory air by a Hans Rudolph mask and direct analysis using an ergospirometer system. The direct gas measurements require expensive and sophisticated equipment as well as trained personnel to perform the test, and this is not standard in many of the out-patient clinics. Thus, the indirect test is cheaper and less time-consuming for the participant and the health personnel making it a more accessible test of cardiorespiratory fitness than the directly measured gas exchange. The indirect estimate of physical performance has, to our knowledge, not yet been validated against the direct gas measurement using the modified Balke protocol in patients with SpA.

Hypothesis and research question The investigators hypothesise that the estimated VO2peak from the maximal CPET is well correlated to the VO2peak measured by direct gas measurements in patients with SpA.

Tests Modified Balke protocol for maximal CPET All participants are asked not to eat for 2-hours prior to the test and to empty their bladder right before the start of measurements. Ahead of the CPET, participants will be familiarised with treadmill walking with a warm-up of 5 minutes at a 1.5% incline. The output setting for the CPET is 4.5% incline and an estimated output level (unfit woman 4.3 km*h-1; unfit man/normal woman 4.7 km*h-1; fit woman/normal man 5.3 km*h-1; fit man 5.3 km*h-1). The incline is increased with 2% every minute, when an incline of 15% is reached the pace of the treadmill is increased with 0.3 km*h-1 every minute while the inclination is kept constant (15%) until participant exhaustion. The test is complete when the participants reach their exhaustion point and are unable to continue the test despite verbal encouragement from the test technician. The protocol is terminated in advance of exhaustion if the test technician observes abnormal and/or adverse test values or the patient requests to stop. Borg RPE ≥ 18, VO2 plateau (two averaged 30-second consecutive measures), age and gender specific reference values for respiratory exchange ratio, blood lactate above age references and the maximal heart rate within 90% of the age-predicted maximum (211-(0.64*age) are used to validate the CPET as a maximal CPET at test termination. Participants who do not fulfil at least 2 of the 4 requirements will be excluded from analyses.

Calculations

For the indirect estimates the maximal CPET data TTE, inclination, and speed is used for calculations of VO2peak. There will use two equations for indirect calculations:

The ACSM equation:

VO2peak = (0.1 * speed (m*s-1) + (1.8 * speed(m*s-1) * inclination (%)) + 3.5

The HUNT3 equation:

Men: 24.24 + (0.599 * inclination) + (3.97 * speed) - (0.122 * body weight) - (0.126 * age) Women: 17.21 + (0.582 * inclination) + (3.317 * speed) - (0.116 * body weight) - (0.099 * age) The two formulas will be compared and validate these calculations against the direct CPET and the non-exercise formula from Kondiskalkulatoren (World Fitness Level).

Measurements The CPET will be performed on a treadmill with 12-lead ECG and scaled by the modified Borg RPE (6-20). Blood pressure is measured before test start (mmHg) and every other minute throughout the test. Heart rate is measured continuously during the CPET and Borg RPE is reported every minute. HRpeak is registered together with the time point of its occurrence. Before the CPET height (m), body weight (kg) and circumference of hip (cm) and waist (cm) are measured. Body composition is measured by bioelectrical impedance analysis (BIA).

Pulmonary function will be assessed by spirometer according to guidelines, and forced expiratory volume (FEV1 L), forced vital capacity (L) and peak expiratory flow (L/min) will be recorded from three attempts at maximal expiratory flow volume loops. Maximal voluntary ventilation (MVV, L/min) will be measured twice by breathing deeply and rapidly for 12 seconds. In cases of poor technique, MVV will be estimated as FEV1 * 37.5. Gas exchange is measured through a Hans Rudolph two-way mask using a breath-by-breath gas analysing system. VO2max is defined as the plateau VO2 of two 30-second samples and the VO2peak is defined as the highest VO2 measured during the test.

Blood lactate concentration is measured in a small blood sample from the fingertip within 60 seconds of test completion to evaluate level of anaerobic processes. CRP is measured in a small blood sample from the fingertip before the CPET for ASDAS calculations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18-70 years old with axial SpA according to ASAS criteria

Exclusion Criteria:

* The American College of Sports Medicine (ACSM) have listed the following contradictions to CPET and participants with absolute or relative contradictions will be excluded.

  * Absolute contraindications to max CPET: acute myocardial infarction within 2 days, unstable angina, uncontrolled cardiac arrhythmia with hemodynamic compromise, active endocarditis, symptomatic severe aortic stenosis, decompensated heart failure, acute pulmonary embolism, pulmonary infarction, or deep venous thrombosis, acute myocarditis or pericarditis, suspected or known aneurysm, acute systemic infection accompanied by fever, body aches, or swollen lymph glands.
  * Relative contraindications to max CPET: Left main coronary stenosis, moderate to severe aortic stenosis, arrhythmia (tachydysrhythmia or bradyarrhythmia), recent stroke or transient ischemic attack, resting hypertension with blood pressure systolic > 200 mmHg and/or diastolic > 115 mmHg, uncorrected medical conditions, such as significant anaemia, important electrolyte abnormalities imbalance, and hyperthyroidism, uncontrolled metabolic disease (e.g. diabetes, thyrotoxicosis or myxoedema) and chronic infectious disease (e.g. mononucleosis, hepatitis, AIDS).
* For the SpA population we have included the following specific exclusion criteria: Unable to walk for less than 15 minutes without support, pregnancy, active uveitis, under- or overweight (BMI: ≤ 18.5 or > 40)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with spondylarthritis diagnosed by a rheumatologist
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-07-09 (Actual); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between VO2peak direct gas measurement and estimated VO2peak ml/minute/kilogram using the modified Balke protocol | 2 hours
  Comparison between the gold standard measurement og cardiorespiratory fitness and the indirect measurements.

SECONDARY OUTCOMES:
Correlation coefficient between VO2peak direct gas measurement and estimated VO2peak ml/minute using the modified Balke protocol | 2 hours
  Comparison between the gold standard measurement og cardiorespiratory fitness and the indirect measurements - not weight adjusted
Performance validation criteria | 2 hours
  To ensure that the participants have performed to their maximal capacity the Borg RPE will be evaluated.
Performance validation criteria | 2 hours
  To ensure that the participants have performed to their maximal capacity the maximal pulse will be evaluated.
Performance validation criteria | 2 hours
  To ensure that the participants have performed to their maximal capacity the lactate level will be evaluated.
Performance validation criteria | 2 hours
  To ensure that the participants have performed to their maximal capacity the expiratory exchange ratio will be evaluated.
Testing non-exercise calculation of physical fitness and two different formulas for indirect calculations | 2 hours
  The HUNT calculations a gender specific, and will be compared to the ACSM calculations Men: 24.24 + (0.599 * inclination) + (3.97 * speed) - (0.122 * body weight) - (0.126 * age) Women: 17.21 + (0.582 * inclination) + (3.317 * speed) - (0.116 * body weight) - (0.099 * age)
Testing non-exercise calculation of physical fitness and two different formulas for indirect calculations | 2 hours
  The ACSM calculation will be compared to the HUNT calculation
Safety measures | 2 hours
  electro cardiogram will be performed prior to and during the exercise test to assess cardiac ischemia (T wave inversion og ST depression > 2 mm) or pathological arrythmia (blockage)
Safety measures | 2 hours
  blood pressure will be performed prior to and during the exercise test to observe for malignant hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte Nellemann, MD PhD, Principal Investigator — Diakonhjemmet Hospital
Locations (1):
- Diakonhjemmet hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No